CLINICAL TRIAL: NCT04153864
Title: Scaling Up Maternal Mental Healthcare by Increasing Access to Treatment (SUMMIT): A Pragmatic, Non-inferiority Trial for Perinatal Depression and Anxiety
Brief Title: Scaling Up Maternal Mental Healthcare by Increasing Access to Treatment (SUMMIT)
Acronym: SUMMIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mount Sinai Hospital, Canada (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Endeavor Health (Other); Women's College Hospital (Other); Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); University of Colorado, Boulder (Other); Harvard Medical School (HMS and HSDM) (Other); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: PCS-2018C1-10621
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Results first posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-07

CONDITIONS: Perinatal Depression
Keywords: Depression; Anxiety; Maternal mental health; Behavioral Activation
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: The intervention modules include:
  1. Brief BA psychological treatment delivered by a non-specialist provider
  2. Brief BA psychological treatment delivered through telemedicine
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators and outcome assessors are independent from type of treatment delivery and allocation status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-specialist (Experimental): Trained non-mental health providers (e.g., nurses or midwives) with general healthcare professional skills (as assessed during recruitment) with no previous experience delivering psychological treatments implementing a brief, manualized behavioral activation treatment
  Interventions: Behavioral: Brief Behavioral Activation Treatment
- Specialist (Active Comparator): Psychiatrists, psychologists and social workers with experience in treating perinatal mental illness and a minimum of 5 years of experience delivering psychological treatments delivering a brief, manualized behavioral activation treatment
  Interventions: Behavioral: Brief Behavioral Activation Treatment
- Telemedicine (Experimental): A brief, manualized behavioral activation treatment delivered over Zoom™ in Toronto, via Webex™ in Chapel Hill, and via Zoom™ in NorthShore
  Interventions: Behavioral: Brief Behavioral Activation Treatment
- In-Person (Active Comparator): A brief, manualized behavioral activation treatment delivered in-person held at participating clinical care sites within UToronto, UNC and NorthShore
  Interventions: Behavioral: Brief Behavioral Activation Treatment

INTERVENTIONS:
Behavioral: Brief Behavioral Activation Treatment — A manualized 6-8 session BA treatment delivered individually to each participant.
  Other Names: Brief evidence-based Psychological Treatment of BA for perinatal depressive and anxiety symptoms

SUMMARY:
SUMMIT's (Scaling Up Maternal Mental health care by Increasing access to Treatment) overarching goal is to examine the scalability and patient-centered provision of brief, evidence-based psychological treatments for perinatal depression and anxiety (N=1226). Specifically, and through a multi-site, randomized, pragmatic trial, the trial examines whether a brief, behavioral activation (BA) treatment delivered via telemedicine is as effective as the same treatment delivered in person; and whether BA delivered by non-mental health providers (e.g., nurses), with appropriate training is as effective as when delivered by specialist providers (psychiatrists, psychologists and social workers) in reducing perinatal depressive and anxiety symptoms. The study will be conducted in Toronto, NorthShore University HealthSystem in Evanston and surrounding areas including Chicago, and North Carolina. The trial will also identify relevant underlying implementation processes and determine whether, and to what extent, these strategies work differentially for certain women over others.

DETAILED DESCRIPTION:
Eligible participants are randomly assigned to the same BA treatment for perinatal depressive and anxiety symptoms in one of four arms: 1) In-person specialist; 2) Telemedicine specialist; 3) In-person non-specialist; 4) Telemedicine non-specialist. However, due to the COVID-19 pandemic, recruitment was adjusted as below:

1. March 2020-July 2021: For the duration of the COVID-19 pandemic period participants were only randomized 1:1 to 1) Telemedicine non-specialist; 2) Telemedicine specialist.
2. July 2021 to January 2022: Randomization of participants to all 4 arms resumed, using a raking approach (weight ratio of 3:1 favoring In-Person to Telemedicine), to rebalance the arms.
3. January 2022 to April 2022: In light of the COVID-19 Omicron variant, participants were only randomized 1:1 to 1) Telemedicine non-specialist; 2) Telemedicine specialist.
4. April 2022 to present: Randomization of participants to all 4 arms resumed at all sites (ratio 1:1:1:1) to 1) In-person specialist; 2) Telemedicine specialist; 3) In-person non-specialist; 4) Telemedicine non-specialist. Randomization to all 4 arms will be followed until in-person arms are fully enrolled after which randomization 1:1 to the two telemedicine arms will be followed. A flexible study design was established at each site based on site-specific COVID restrictions.

This approach was verified by the study statistician, an independent methodologist and the study funder. All analyses will be run as both intent-to-treat and per protocol.

ELIGIBILITY:
Inclusion Criteria:

* EPDS≥10
* ≥18 years
* Pregnant up to 36 weeks or 4-30 weeks postpartum
* Speaks English or (US sites) Spanish

Exclusion Criteria:

* Active suicidal intent (ideation and plan), active symptoms of psychosis or mania
* Psychotropic medication dose or medication change within two weeks of enrollment or beginning treatment
* Ongoing psychotherapy (no more than once every 8 weeks or during the duration of the intervention)
* Active substance abuse or dependence
* Severe fetal anomalies, stillbirth or infant death at time of enrollment for index pregnancy
* Non-English, non-Spanish speakers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1230 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2024-02-26 (Actual); Study Completion 2025-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daisy R Singla, PhD, Principal Investigator — Sinai Health System
Locations (5):
- United States (2):
  - NorthShore University Health System, Evanston, Illinois
  - University of North Carolina, Chapel Hill, North Carolina
- Canada (3):
  - St. Michael's Hospital, Toronto, Ontario
  - Sinai Health System, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Bradley RH, Caldwell BM. The HOME Inventory and family demographics. Developmental Psychology 1984; 20(2): 315.
- [Background] Bayley N. Bayley Scales of Infant Development and Toddler Development: Technical Manual: The PsychCorp; 2006.
- [Background] McCabe-Beane JE, Segre LS, Perkhounkova Y, Stuart S, O'Hara MW. The identification of severity ranges for the Edinburgh Postnatal Depression Scale. Journal of Reproductive and Infant Psychology. 2016;34(3):293-303.
- [Background] Simpson W, Glazer M, Michalski N, Steiner M, Frey BN. Comparative efficacy of the generalized anxiety disorder 7-item scale and the Edinburgh Postnatal Depression Scale as screening tools for generalized anxiety disorder in pregnancy and the postpartum period. Can J Psychiatry. 2014 Aug;59(8):434-40. doi: 10.1177/070674371405900806. PMID 25161068
- [Derived] Andrejek N, Lea Z, Cussons A, Sandeep S, Dennis CL, La Porte LM, Vigod SN, Silver RK, Meltzer-Brody S, Singla DR. Advancing telemedicine and task-sharing to improve access to psychotherapy for perinatal populations. Commun Med (Lond). 2025 Sep 30;5(1):406. doi: 10.1038/s43856-025-01099-9. PMID 41028222
- [Derived] Zaidan M, Lawson AS, Andrejek N, Walsh K, Dennis CL, Meltzer-Brody S, Silver RK, Stuebe AM, Vigod SN, Singla DR. Bridges to treatment satisfaction: the roles of trauma, social support, race and ethnicity among perinatal women receiving behavioural activation therapy. BMC Med. 2025 Aug 20;23(1):489. doi: 10.1186/s12916-025-04272-y. PMID 40835941
- [Derived] Kaliush PR, Molina NC, Berenbaum TS, Dennis CL, Gaynes BN, Meltzer-Brody S, Reyes-Rodriguez ML, Silver RK, Stuebe AM, Vigod SN, Schiller CE, Singla DR. Behavioral Activation for Perinatal Suicide Ideation: Secondary Analysis of a Noninferiority Randomized Clinical Trial. JAMA Psychiatry. 2025 Dec 1;82(12):1234-1239. doi: 10.1001/jamapsychiatry.2025.2116. PMID 40833774
- [Derived] Singla DR, Silver RK, Vigod SN, Schoueri-Mychasiw N, Kim JJ, La Porte LM, Ravitz P, Schiller CE, Lawson AS, Kiss A, Hollon SD, Dennis CL, Berenbaum TS, Krohn HA, Gibori JE, Charlebois J, Clark DM, Dalfen AK, Davis W, Gaynes BN, Leszcz M, Katz SR, Murphy KE, Naslund JA, Reyes-Rodriguez ML, Stuebe AM, Zlobin C, Mulsant BH, Patel V, Meltzer-Brody S. Task-sharing and telemedicine delivery of psychotherapy to treat perinatal depression: a pragmatic, noninferiority randomized trial. Nat Med. 2025 Apr;31(4):1214-1224. doi: 10.1038/s41591-024-03482-w. Epub 2025 Mar 3. PMID 40033113
- [Derived] Singla DR, Hossain S, Andrejek N, Cohen MJ, Dennis CL, Kim J, La Porte L, Meltzer-Brody SE, Puerto Nino A, Ravitz P, Schoueri-Mychasiw N, Silver R, Vigod SN, Zibaman M, Schiller CE. Culturally sensitive psychotherapy for perinatal women: A mixed methods study. J Consult Clin Psychol. 2022 Oct;90(10):770-786. doi: 10.1037/ccp0000754. Epub 2022 Sep 29. PMID 36174135
- [Derived] Singla DR, Meltzer-Brody SE, Silver RK, Vigod SN, Kim JJ, La Porte LM, Ravitz P, Schiller CE, Schoueri-Mychasiw N, Hollon SD, Kiss A, Clark D, Dalfen AK, Dimidjian S, Gaynes BN, Katz SR, Lawson A, Leszcz M, Maunder RG, Mulsant BH, Murphy KE, Naslund JA, Reyes-Rodriguez ML, Stuebe AM, Dennis CL, Patel V. Scaling Up Maternal Mental healthcare by Increasing access to Treatment (SUMMIT) through non-specialist providers and telemedicine: a study protocol for a non-inferiority randomized controlled trial. Trials. 2021 Mar 5;22(1):186. doi: 10.1186/s13063-021-05075-1. PMID 33673867

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from January 2020 to October 2023 from five clinical sites (Mount Sinai Hospital, Women's College Hospital, St. Michael's Hospital, University of North Carolina and Endeavor Health).
Pre-assignment Details: A total of 3,629 individuals were approached. 1,543 agreed to participate by completing the consent form and 1,512 completed a second, more detailed screening. A total of 1,230 participants were enrolled and randomized into the trial.
Groups:
- Arm 1: Telemedicine Non-Specialist: The participants in this group were randomly assigned to receive Telemedicine, with a Non-Specialist provider.
- Arm 2: In-Person Non-Specialist: The participants in this group were randomly assigned to receive In-Person care, with a Non-Specialist provider
- Arm 3: Telemedicine Specialist: The participants in this group were randomly assigned to receive Telemedicine, with a Specialist provider.
- Arm 4: In-Person Specialist: The participants in this group were randomly assigned to receive In-Person care, with a Specialist provider.
Period: Overall Study
Arm/Group | Arm 1: Telemedicine Non-Specialist | Arm 2: In-Person Non-Specialist | Arm 3: Telemedicine Specialist | Arm 4: In-Person Specialist
Started | 472 | 145 | 469 | 144
Completed (Completion here is defined as trial participants who completed the primary outcome (EPDS) at 3-month follow-up assessment; data from the 6- and 12-month follow-up assessments have been collected and will be published by February 2026) | 419 | 128 | 417 | 134
Not Completed | 53 | 17 | 52 | 10
Not completed — Withdrawal by Subject | 21 | 7 | 23 | 2
Not completed — Lost to Follow-up | 4 | 0 | 3 | 0
Not completed — Did not complete 3-month follow-up assessment but continued in the trial | 28 | 10 | 26 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm 1: Telemedicine Non-Specialist | Arm 2: In-Person Non-Specialist | Arm 3: Telemedicine Specialist | Arm 4: In-Person Specialist | Total
Number analyzed (Participants) | 472 | 145 | 469 | 144 | 1230
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Demographic data is missing for 4 participants, distributed as follows:
  Arm 1 = 1 Arm 3 = 3
  years
    number analyzed (Participants) | 471 | 145 | 466 | 144 | 1226
    (all) | 33.08 (5.10) | 33.84 (4.79) | 33.04 (4.79) | 34.10 (5.01) | 33.27 (4.95)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 441 | 144 | 440 | 143 | 1168
  Different Identity | 1 | 0 | 0 | 0 | 1
  Genderqueer/Gender non-confirming | 2 | 0 | 0 | 0 | 2
  Prefer not to answer | 1 | 0 | 1 | 0 | 2
  Not reported | 27 | 1 | 28 | 1 | 57
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaska Native | 1 | 0 | 3 | 1 | 5
  Asian | 87 | 27 | 73 | 22 | 209
  Black/African American | 40 | 19 | 46 | 19 | 124
  Hawaiian/Pacific Islander | 1 | 1 | 1 | 1 | 4
  White | 242 | 69 | 231 | 72 | 614
  Multi-race | 34 | 10 | 45 | 11 | 100
  Hispanic (Latino/Latina) | 38 | 10 | 39 | 14 | 101
  Other | 15 | 4 | 14 | 2 | 35
  Prefer not to answer | 13 | 5 | 14 | 2 | 34
  Not reported | 1 | 0 | 3 | 0 | 4
Baseline EPDS [Mean (Standard Deviation); unit: units on a scale] — Edinburgh Postnatal Depression Scale (EPDS) is a brief, 10-item self-administered questionnaire used to help identify perinatal depressive symptoms. Each item is scored from 0 to 3, with a total summed score ranging from 0-30. Higher EPDS total scores indicates higher severity of depressive symptoms.
  units on a scale | 15.63 (3.76) | 15.68 (3.83) | 15.96 (3.92) | 15.72 (3.96) | 15.77 (3.85)
Baseline GAD-7 [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder (GAD-7) is a brief, 7-item self-administered questionnaire used to screen for and assess the anxiety symptoms. Each item is scored from 0 to 3, with a total summed score ranging from 0-21. Higher GAD-7 total scores indicates a greater severity of anxiety symptoms.
  units on a scale | 11.92 (4.76) | 12.00 (4.54) | 11.72 (5.11) | 11.87 (5.08) | 11.85 (4.90)

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms: Edinburgh Postnatal Depression Scale (EPDS) Mean Score
Description: Edinburgh Postnatal Depression Scale (EPDS) is a brief, 10-item self-administered questionnaire used to help identify perinatal depressive symptoms. Each item is scored from 0 to 3, with a total summed score ranging from 0-30. Higher EPDS total scores indicates higher severity of depressive symptoms.
Time Frame: 3-months post-randomization
Population: 1. The groups shown below are non-mutually exclusive, as participants were included in two arms (as reflected in the four arms described in the Participant Flow table). This overlap occurred because the study used a 2 × 2 factorial design, in which participants simultaneously received a combination of two interventions.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- Non-Specialist: Trained non-mental health providers (e.g., registered nurses, midwives and doulas) without formal training in mental health care or previous experience delivering psychological treatments.
- Specialist: Psychiatrists, psychologists and social workers with a minimum of 5 years of experience delivering psychological treatments delivering a brief, manualized behavioral activation treatment
- Telemedicine: A brief, manualized behavioral activation treatment delivered over a secure HIPPA/PHIPPA compliant audio-visual digital platform (i.e., Zoom™ in Toronto, via Webex™ in Chapel Hill, and via Zoom™ in Chicago)
- In-Person: A brief, manualized behavioral activation treatment delivered in-person held at participating clinical care sites within Toronto, Chapel Hill and Chicago
Arm/Group | Non-Specialist | Specialist | Telemedicine | In-Person
Number analyzed (Participants) | 547 | 551 | 836 | 262
score on a scale | 9.27 [8.85 to 9.70] | 8.91 [8.49 to 9.33] | 9.15 [8.79 to 9.50] | 8.92 [8.38 to 9.45]
Statistical Analysis 1: Comparison: Non-Specialist vs Specialist; Behavioral Activation (BA) delivered by Non-Specialists will be non-inferior to BA delivered by Specialists if the upper limit of the 95% confidence interval for the estimated mean difference in EPDS scores is less than the pre-specified 10% non-inferiority margin (NIM); Test type: Non-Inferiority — The Non-Inferiority Margin (NIM) was defined as 10% of the mean EPDS score in the Specialist group (8.91), which corresponded to a value of 0.89. This predetermined NIM of 10% aligns with noninferiority guidelines and ensures clinically meaningful conclusions; p < 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.36, 95% CI 1-sided [upper limit 0.86]
Statistical Analysis 2: Comparison: Telemedicine vs In-Person; Behavioral Activation (BA) delivered via Telemedicine will be non-inferior to BA delivered In-Person if the upper limit of the 95% confidence interval for the estimated mean difference in EPDS scores is less than the pre-specified 13% non-inferiority margin (NIM). Please note, this presents the Intention to Treat (ITT) analysis; Test type: Non-Inferiority — The NIM was defined as 13% of the mean EPDS score in the In-Person group (8.92), which corresponded to a value of 1.16. This predetermined NIM of 13% aligns with noninferiority guidelines and ensures clinically meaningful conclusions; p < 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.23, 95% CI 1-sided [upper limit 0.77]
Statistical Analysis 3: Comparison: Telemedicine vs In-Person; Behavioral Activation (BA) delivered via Telemedicine will be non-inferior to BA delivered In-Person if the upper limit of the 95% confidence interval for the estimated mean difference in EPDS scores is less than the pre-specified 13% non-inferiority margin (NIM). Please note, this is per protocol analysis. Due to institutional pandemic-related restrictions, 21 participants were switched from In-Person to Telemedicine and met criteria for the per protocol analyses; Test type: Non-Inferiority — The NIM was defined as 13% of the mean EPDS score in the In-Person group (8.81), which corresponded to a value of 1.15. This predetermined NIM of 13% aligns with noninferiority guidelines and ensures clinically meaningful conclusions; p < 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.36, 95% CI 1-sided [upper limit 0.91]

2. Secondary Outcome: Depressive Symptoms: Edinburgh Postnatal Depression Scale (EPDS) Mean Score
Description: as for outcome 1
Time Frame: 6- and 12-months post-randomization
Reporting Status: Not Posted

3. Secondary Outcome: Anxiety Symptoms: Generalized Anxiety Disorder Scale (GAD-7) Mean Score
Description: Generalized Anxiety Disorder (GAD-7) is a brief, 7-item self-administered questionnaire used to screen for and assess the anxiety symptoms. Each item is scored from 0 to 3, with a total summed score ranging from 0-21. Higher GAD-7 total scores indicates a greater severity of anxiety symptoms.
Time Frame: 3-months post-randomization
Population: 1. The groups shown below are non-mutually exclusive, as participants were included in two arms (the four arms described in the Participant Flow table). This overlap occurred because the study used a 2 × 2 factorial design, in which participants simultaneously received combinations of two interventions.
  2. At 3-months post-randomization, GAD-7 data were missing for some participants; the numbers presented above reflect only those with available data and used for analysis.
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Non-Specialist | Specialist | Telemedicine | In-Person
Number analyzed (Participants) | 545 | 550 | 834 | 261
units on a scale | 6.44 [6.01 to 6.86] | 6.36 [5.95 to 6.78] | 6.43 [6.09 to 6.78] | 6.29 [5.71 to 6.88]
Statistical Analysis 1: Comparison: Non-Specialist vs Specialist; Behavioral Activation (BA) delivered by Non-Specialists will be non-inferior to BA delivered by Specialists if the upper limit of the 95% confidence interval for the estimated mean difference in GAD-7 scores is less than the pre-specified 10% non-inferiority margin (NIM).This analysis was performed on 3-months post-randomization scores; Test type: Non-Inferiority — The NIM was defined as 10% of the mean GAD-7 score for the Specialist group (6.36), which corresponded to a value of 0.64. This predetermined NIM of 10% aligns with noninferiority guidelines and ensures clinically meaningful conclusions; p < 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.08, 95% CI 1-sided [upper limit 0.57]
Statistical Analysis 2: Comparison: Telemedicine vs In-Person; Behavioral Activation (BA) delivered via Telemedicine will be non-inferior to BA delivered In-Person if the upper limit of the 95% confidence interval for the estimated mean difference in GAD-7 scores is less than the pre-specified 13% non-inferiority margin (NIM). Please note, this presents the Intention to Treat (ITT) analysis; Test type: Non-Inferiority — The NIM was defined as 13% of the mean GAD-7 score in the In-Person group (6.29), which corresponded to a value of 0.82. This predetermined NIM of 13% aligns with noninferiority guidelines and ensures clinically meaningful conclusions; p < 0.05, t-test, 1 sided; Mean Difference (Final Values) = 0.14, 95% CI 1-sided [upper limit 0.73]

4. Secondary Outcome: Child Mental Health Development
Description: Child mental development was measured by Bayley Mental Developmental Scale IV and the provision of psychosocial stimulation by the mother (study participant) as measured by the Home Observation Measurement Evaluation. The Bayley Mental Developmental Scale IV was used to measure cognitive development and expressive and receptive language in participants' children. The composite scores are scaled to a metric, with a mean of 100, standard deviation of 15, and range of 40 to 160. Higher scaled scores are associated with higher mental health development in children. The minimum and maximum values for the Home Observation Measurement Evaluation scale scores are 0 and 45 respectively. Higher scores are associated with a more enriched environment.
Time Frame: 6 to 24 months post child birth (extended due to COVID-19)
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Baseline to 3-months post-randomization
Description: We reported all Serious Adverse Events (SAEs) to the Data Safety Monitoring Board (DSMB) within 72 hours of a confirmed SAE. We reported all Adverse Events (AEs) to the DSMB within 5 days of a confirmed AE as per the study's safety protocols and DSMB charter.
Groups:
- Arm 4: In-Person Specialist (4): The participants in this group were randomly assigned to receive In-Person care, with a Specialist provider.
Arm/Group | Arm 1: Telemedicine Non-Specialist | Arm 2: In-Person Non-Specialist | Arm 3: Telemedicine Specialist | Arm 4: In-Person Specialist (4)
All-Cause Mortality (participants affected / at risk) | 1/472 | 0/145 | 0/469 | 0/144
Serious Adverse Events (participants affected / at risk) | 10/472 | 2/145 | 6/469 | 0/144
Other Adverse Events (participants affected / at risk) | 1/472 | 0/145 | 0/469 | 1/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Telemedicine Non-Specialist (N=472) | Arm 2: In-Person Non-Specialist (N=145) | Arm 3: Telemedicine Specialist (N=469) | Arm 4: In-Person Specialist (4) (N=144)
Fetal or infant death (General disorders) | 5 | 0 | 1 | 0
Hospitalization (General disorders) | 1 | 1 | 3 | 0
Life threatening events in the mother, fetus, neonate or infant (General disorders) | 1 | 0 | 0 | 0
Maternal death (General disorders) | 1 | 0 | 0 | 0
Other serious important medical events (General disorders) | 1 | 0 | 1 | 0
Hospitalization + Life threatening events in the mother, fetus, neonate or infant (General disorders) | 1 | 1 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Telemedicine Non-Specialist (N=472) | Arm 2: In-Person Non-Specialist (N=145) | Arm 3: Telemedicine Specialist (N=469) | Arm 4: In-Person Specialist (4) (N=144)
Imminent and active suicidal intent (Psychiatric disorders) | 0 | 0 | 0 | 1
Increase in depressive symptoms (Psychiatric disorders) | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-10-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04153864/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-16): https://cdn.clinicaltrials.gov/large-docs/64/NCT04153864/SAP_001.pdf